CLINICAL TRIAL: NCT01447108
Title: Examining the Efficacy of Low Intensity Low Frequency Surface Acoustic Wave Ultrasound(LILF/SAWU) in Trigeminal Neuralgia Pain
Brief Title: Surface Acoustic Wave Ultrasound in Trigeminal Neuralgia Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Manuel Zwecker MD, Senour physician at the Department of Neurological Rehabilitation, Sheba Medical Center
Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-8601-11-MZ-CTIL
Record Dates: First submitted 2011-09-15; First posted 2011-10-05 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Trigeminal Neuralgia; Tic Douloureux
Keywords: Trigeminal Neuralgia; Tic Douloureux; Low Intensity Low Frequency Surface Acoustic Wave Ultrasound
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- TN patients (Experimental): Patients suffering from Trigeminal neuralgia
  Interventions: Device: Low Intensity Low Frequency Surface Acoustic Wave Ultrasound (PainShield™)

INTERVENTIONS:
Device: Low Intensity Low Frequency Surface Acoustic Wave Ultrasound (PainShield™) — All subjects will be treated four weeks with a placebo PainShield™ while continuing with their current pharmaco- analgesic regimen. Aferterwards all subjects will be crossed over to active Painshield™ therapy for the next four weeks.
  The Painshield™ device is a patch, which will be applied to their forehead for six-eight hours during night while sleeping.
  Other Names: PainShield™

SUMMARY:
The "Suicide Disease", Trigeminal Neuralgia (TN) is arguably caused by one of the most discrete and eloquently reversible central nervous system lesions known to the field of neurology.

Recently Dr Adahan H. and Dr Binshtok A. have completed an open label series of 25 subjects with refractory TN showing a remarkable positive response rate to TN's treatment with Low Intensity Low Frequency Surface Acoustic Wave Ultrasound (LILF/SAWU).

The primary objective of this study, therefore, is to determine whether this apparent efficacy of Low Intensity Low Frequency Ultrasound (LILFU) in the treatment of TN pain could withstand the rigors of an n=1 crossover placebo control study.

Participants with refractory trigeminal neuralgia pain despite optimized pharmacotherapy for at least six months will be screened for participation in the study based on rigorous inclusion and exclusion criteria. It is judged rather unlikely that such subjects will experience spontaneous regression of their disease in the course of this study.

Patients meeting the inclusion criteria will be treated with four weeks of a placebo Low Intensity Low Frequency Surface Acoustic Wave Ultrasound (LILF/SAWU) device while continuing with their pharmaco-analgesic regimen. All patients will be crossed over to active LILF/SAWU therapy for the next four weeks. Patients will be blinded to all treatments throughout the study. Patients will be instructed to use the device daily overnight, and remove it upon wakening. The device is programmed to work in cycles of 30 minutes on and 30 minutes off, for a total of six- eight hours of intermittent treatment.

At the end of the second month of the study, patients will be offered a choice as to whether they wished to continue with the current (active) device or go back to the 1st (sham) device.

Patient's pain severity will be tracked every two weeks over the course of three months. Functional health and well being will be monitored at intake, post "Placebo" period, post "Active" period and at completion of the study.

DETAILED DESCRIPTION:
1. Introduction:

   Trigeminal neuralgia (TN) is one of the most severe and progressive forms of chronic neuropathic pain.

   The latest scientific work has shown that the most likely cause of TN is a highly reversible tiny central nervous system (CNS) lesion at the root entry zone (REZ) of the trigeminal nerve measuring less than 0.5 cm cubed.

   The presence of a discrete, highly eloquent and highly reversible central nervous system (CNS) lesion presents a unique opportunity to test and measure the neuroegenerative potential of therapeutic modalities that can be effectively delivered to the site of this pathology.

   Ultrasound has been shown to be an effective treatment for the demyelination found in carpal tunnel syndrome in man ( Ebenbicher , Resch , Nicolakis, Weisinger ,Uhl, Ghanemm and Fialka 1998) , with numerous research studies showing its ability to accelerate peripheral nerve regeneration and functional recovery in rats(Crisci and Ferreria, 2002). There is also a growing body of scientific evidence demonstrating the efficacy of ultrasound in facilitating wound healing and analgesia. Numerous published research studies of ultrasound, and specifically LILFU, have provided Level 1 evidence of efficacy in bone healing, prevention and treatment of fracture non-union, acceleration of fracture healing, and it is also showing promise in the field of tendon healing. (Campbell C.K and Jorns 2007). In vitro, low-intensity ultrasound, has been shown to have direct non thermal effects on cell physiology, stimulating the expression of numerous genes involved in the healing process, including aggrecan, an insulin-like growth factor, transforming collagen, nitric oxide synthase, cytokines, and angiogenesis (Devor, Amir and Rappaport , 2002).

   A dynamic balance appears to exist between ongoing neural damage from the repetitive mechanical stress at the sight of neurovascular compression and the ongoing efforts of the LILFU to repair the damage via endogenous remyelination. The investigators hypothesize that the nature of this balance may determine whether the TN sufferer finds himself in either a TN pain crisis or remission. This would explain the remission recurrence pattern typically seen in the early course of the disease as well as the progressive nature of the illness, which may be attributable to the progressive effect of repetitive micro-injury. It is possible that LILF/SAWU might be the catalyst in promoting neuroregeneration thus helping induce and sustain remission
2. Rationale of the study TN, a form of neuropathic pain, is generally considered one of the most severe and life disrupting pains known to patients. Unfortunately, in most people, TN is a progressive illness that intensifies and becomes more difficult to control over the years. Medication, although often initially affective, usually loses its effectiveness over the trajectory course of the illness. Each patient with TN has a different response to these medications and to his/her pain, but over the years of disease progression, many will eventually find that medications do not adequately control their progressively worsening condition. (Zakrezewska and Linskey, 2009) Medication has not been shown to slow the progression of the disease. On the contrary, over the years, many people find themselves having to take higher doses of medication or having to take several different medications together to control their pain with a resultant accumulation of problematic side effects. Eventually, over the long term, more than half of trigeminal neuralgia patients will seek a surgical solution to manage their pain.(Zakrezewska et al.2009) There is a growing emphasis and desire for minimally invasive therapy and treatments of all abnormal pathologies and disease particularly TN. Although stereotactic radio-surgery is presently one of the least invasive procedures, it does have some potentially serious adverse effect, such as permanent nerve damage, causing weakness and sensory impairment, and in some cases anesthesia dolorosa, which can also occur with all ablative procedures (Emril and Ho, 2010) As stated earlier, this intractable pain appears due to a highly reversible micro lesion in the CNS at the REZ of the trigeminal nerve is considered to be the result of focal microvascular compression. The resulting demyelination and dysmyelination contributes to ephatic transmission between large myelinated fibers and pain conducting C-fibers possibly triggered by the pulsatile compression of the artery against the injured nerve. The reversibility of this small CNS injury is witnessed by the rapid onset of recovery of Somatosensory Evoked Potentials (SSEP's) measured pre-operatively at the time of surgical decompression as well as by the fact that anatomical studies show little axon-notmesis.( Leandri 2002 , Devor 2002 and Love, 1998) ) Our hypothesis is that the initial intermittent nature of TN pain is witness to the delicate balance between repetitive injury to the REZ of the trigeminal nerve and the bodies inherent ability to overcome it as shown by anatomical studies showing signs of remyelination. The presence of a discrete yet highly reversible CNS lesion presents a unique opportunity for our future research to test and objectively measure the neuroregenerative potential of therapeutic modalities that can be effectively delivered to the site of this pathology in an attempt to reinforce the potential of the CNS to regenerate the CNS myelin destroyed by this disease.

   Today, there are no readily accessible therapies for central or peripheral neuropathic pain that hold the promise of facilitating neuroregeneration.

   Ultrasound delivered to injured nerves has been shown in five animal studies in the past eight years to have neuroregenerative capacities and has also been associated with improved remyelination in carpal tunnel syndrome in humans in one RCT (Ebenbicher , Resch , Nicolakis, Weisinger ,Uhl, Ghanemm and Fialka 1998) Ultrasound delivered to injured nerves has been shown in several studies to reverse nerve damage commonly seen in the trigeminal nerve of patient's with TN.(Crisci 2002, Chang 2004, Mourad 2001, Paik 2002, Zhou 2006) Traditional high energy, high frequency bulk wave ultrasound devices does not penetrate the cranium and cannot, therefore, be used for treating the REZ of the trigeminal ganglion. Until the advent of the Painshield™ device, low intensity, low frequency surface acoustic wave ultrasound technology (LILF/SAWU) had not been applied in the field of medicine. It is, however, ever-present in cell phone devices' electronic circuits (Campell C.K). Based on the known physical properties of SAW acoustics, it is expected that when a SAW transducer is applied to a surface which has underlying bone, such as the forehead, the energy spreads over the entire surface of the bony skull and its internal foramina. It is efficiently transmitted via the cerebrospinal fluid (CSF) to the CNS structures situated close to or beside the bony structures. Hence, the REZ and ganglion of the trigeminal nerve, as well as the entire length of all its branches, are exposed to potentially healing acoustic ultrasound energy.

   The PainShieldTM system is a novel, patch based therapeutic ultrasound product, Food and Drug Administration (FDA) approved for the treatment of painful conditions, including trigeminal neuralgia. The device is a portable and battery powered and can be connected to a disposable patch through which it delivers localized energy creating waves, which affect localized pain and induce soft tissue healing. This is made possible due to the company's proprietary technology which allows for the creation of a therapeutic transducer that can be made disposable and incorporated into a patch. Until the Painshield™ technology came to light; there was no available ultrasound device that could safely deliver surface acoustic ultrasound technology intracranially, for up to several hours daily.

   In this single blinded crossover study, the investigators aim to determine the effectiveness of Low Intensity Low Frequency Surface Acoustic Wave Ultrasound (LILF/SAWU) in the treatment of TN pain.
3. Objectives and Hypothesis:

   The primary objective of this study is to determine the effectiveness of Low Intensity Low Frequency Ultrasound Surface Acoustic Wave (LILFU/SAW) in the treatment of TN using a single blind n=1 cross over study design.

   Our hypothesis (H1) is that LILFU treatment, via Painshield™, will provide pain relief in patients suffering with chronic TN as measured by the modified Barrow Neurological Index score.

   The investigators further hypothesize (H2) that following this relief in pain the TN sufferers will enjoy improved functional health and well being as measured by the SF-36.

   This in turn will lead to a further hypothesis (H3) that the TN sufferers will reduce the amount of medication they consume each month, as reported by the participants themselves.
4. Study Design:

The study is designed as a single blind crossover trial. This design was chosen because TN is a rare disease and recruitment of adequate subjects for a formal RCT would prove too difficult. Subjects diagnosed with refractory TN for at least six months despite currently undergoing optimized pharmacotherapy (BNI V) will be treated with four weeks of a placebo PainSheield™ while continuing with their current pharmaco- analgesic regimen. All patients will be crossed over to active Painshield™ therapy for the next four weeks. They will apply the Painshield™ patch to their forehead for six-eight hours a night (depends on how many hours they sleep) for the four weeks.

At the end of the second month of the study, patients will be offered to either continue with active PainShield™ treatment for the third and final month, or return to the "sham" PainShield™ treatment.

Assessment of pain via the BNI index and Short form MCGILL Pain Questionnaire ("SFMPQ") will be recorded at two week intervals throughout the three months of the study. Functional health and wellbeing will be measured by the SF-36 Questionnaire at intake, cross over time (initial four weeks), post "Active" treatment and at the end of the three month study period.

Statistical Analysis:

The following parameters will be calculated:

1. Mean scores of the Barrow Neurological Index.
2. Mean scores for each SF-36 dimensions (General health, role limitation due to a physical problem, physical function and bodily pain).
3. Percentage of patients who chose to continue with the active Painshield™ treatment for further four weeks.
4. Proportion/ percentage of BNI scores- Initial response to treatment will be defined as an improvement in patient-reported BNI score to a level of BNI< IIIB.

Comparisons of BNI scores between groups will be evaluated using following statistical tests: independent paired T-test for SF-36 scores, Wilcoxon test for BNI scores, and Chi-Square test in order to calculate the proportion of BNI scores.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with trigeminal neuralgia refractory to medical treatment (modified BNI V).

Exclusion Criteria:

* Male or female, under the age of 18.
* Active illicit drug use
* Pregnancy.
* Psychiatric illness which may prevent the patient from participation in the study.
* Anesthesia dolorosa with pain greater than or equal to 3/10
* Dental implants.
* Other known pathology of the trigeminal nerve including iatrogenic anesthesia dolorosa.
* Cancer and bone metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Level of pain | Change in level of pain from baseline to after two months of treatment
  Barrow Neurological Index score (BNI ) pain intensity scale will be used
Pain intensity and quality of pain | Change in intensity and quality of pain from baseline to after two months of treatment
  "SFMPQ" - Short form MCGILL Pain Questionnaire will be used.
Functional Health and Wellbeing | Change in functional health and wellbeing from baseline to after two months of treatment
  SF-36 Questionnaire will be used

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Zwecker, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Crisci AR, Ferreira AL. Low-intensity pulsed ultrasound accelerates the regeneration of the sciatic nerve after neurotomy in rats. Ultrasound Med Biol. 2002 Oct;28(10):1335-41. doi: 10.1016/s0301-5629(02)00576-8. PMID 12467860
- [Background] Chang CJ, Hsu SH. The effects of low-intensity ultrasound on peripheral nerve regeneration in poly(DL-lactic acid-co-glycolic acid) conduits seeded with Schwann cells. Ultrasound Med Biol. 2004 Aug;30(8):1079-84. doi: 10.1016/j.ultrasmedbio.2004.06.005. PMID 15474752
- [Background] Mourad PD, Lazar DA, Curra FP, Mohr BC, Andrus KC, Avellino AM, McNutt LD, Crum LA, Kliot M. Ultrasound accelerates functional recovery after peripheral nerve damage. Neurosurgery. 2001 May;48(5):1136-40; discussion 1140-1. doi: 10.1097/00006123-200105000-00035. PMID 11334281
- [Background] Paik NJ, Cho SH, Han TR. Ultrasound therapy facilitates the recovery of acute pressure-induced conduction block of the median nerve in rabbits. Muscle Nerve. 2002 Sep;26(3):356-61. doi: 10.1002/mus.10209. PMID 12210364
- [Background] Ebenbichler GR, Resch KL, Nicolakis P, Wiesinger GF, Uhl F, Ghanem AH, Fialka V. Ultrasound treatment for treating the carpal tunnel syndrome: randomised "sham" controlled trial. BMJ. 1998 Mar 7;316(7133):731-5. doi: 10.1136/bmj.316.7133.731. PMID 9529407
- [Background] Campbell C. K. Surface Acoustic wave devices for mobile and wireless communications. Chapter-Fundamentals of surface acoustic waves and devices. Academic press NY p20-25.
- [Background] Jorns TP, Zakrzewska JM. Evidence-based approach to the medical management of trigeminal neuralgia. Br J Neurosurg. 2007 Jun;21(3):253-61. doi: 10.1080/02688690701219175. PMID 17612914
- [Background] Devor M, Amir R, Rappaport ZH. Pathophysiology of trigeminal neuralgia: the ignition hypothesis. Clin J Pain. 2002 Jan-Feb;18(1):4-13. doi: 10.1097/00002508-200201000-00002. PMID 11803297
- [Background] Leandri M, Eldridge P, Miles J. Recovery of nerve conduction following microvascular decompression for trigeminal neuralgia. Neurology. 1998 Dec;51(6):1641-6. doi: 10.1212/wnl.51.6.1641. PMID 9855516
- [Background] Devor M, Govrin-Lippmann R, Rappaport ZH. Mechanism of trigeminal neuralgia: an ultrastructural analysis of trigeminal root specimens obtained during microvascular decompression surgery. J Neurosurg. 2002 Mar;96(3):532-43. doi: 10.3171/jns.2002.96.3.0532. PMID 11883839
- [Background] Love S, Hilton DA, Coakham HB. Central demyelination of the Vth nerve root in trigeminal neuralgia associated with vascular compression. Brain Pathol. 1998 Jan;8(1):1-11; discussion 11-2. doi: 10.1111/j.1750-3639.1998.tb00126.x. PMID 9458161
- [Background] Poole HM, Murphy P, Nurmikko TJ. Development and preliminary validation of the NePIQoL: a quality-of-life measure for neuropathic pain. J Pain Symptom Manage. 2009 Feb;37(2):233-45. doi: 10.1016/j.jpainsymman.2008.01.012. Epub 2008 Aug 3. PMID 18676118
- [Background] Rogers CL, Shetter AG, Fiedler JA, Smith KA, Han PP, Speiser BL. Gamma knife radiosurgery for trigeminal neuralgia: the initial experience of The Barrow Neurological Institute. Int J Radiat Oncol Biol Phys. 2000 Jul 1;47(4):1013-9. doi: 10.1016/s0360-3016(00)00513-7. PMID 10863073
- [Background] Azar M, Yahyavi ST, Bitaraf MA, Gazik FK, Allahverdi M, Shahbazi S, Alikhani M. Gamma knife radiosurgery in patients with trigeminal neuralgia: quality of life, outcomes, and complications. Clin Neurol Neurosurg. 2009 Feb;111(2):174-8. doi: 10.1016/j.clineuro.2008.09.020. Epub 2008 Nov 7. PMID 18995955
- [Background] Lewin-Epstein N, Sagiv-Schifter T, Shabtai EL, Shmueli A. Validation of the 36-item short-form Health Survey (Hebrew version) in the adult population of Israel. Med Care. 1998 Sep;36(9):1361-70. doi: 10.1097/00005650-199809000-00008. PMID 9749659
- [Background] Zakrzewska JM, Linskey ME. Trigeminal neuralgia. BMJ Clin Evid. 2009 Mar 12;2009:1207. PMID 19445753
- [Background] Sarlani E, Balciunas BA, Grace EG. Orofacial pain--Part I: Assessment and management of musculoskeletal and neuropathic causes. AACN Clin Issues. 2005 Jul-Sep;16(3):333-46. doi: 10.1097/00044067-200507000-00007. PMID 16082236
- [Background] Emril DR, Ho KY. Treatment of trigeminal neuralgia: role of radiofrequency ablation. J Pain Res. 2010 Dec 12;3:249-54. doi: 10.2147/JPR.S14455. PMID 21311718